CLINICAL TRIAL: NCT02510898
Title: Examining the Role of Expressive Writing (EW) to Improve Resilience Among Those Experiencing an Emotional Upheaval or a Physical Health Challenge
Brief Title: Examining the Role of Expressive Writing (EW) to Improve Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00062054
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Resilience

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Arm (Experimental): All subjects enrolled in the study will receive the intervention. This is a one-arm study.
  Interventions: Behavioral: 6-week Writing to Heal course

INTERVENTIONS:
Behavioral: 6-week Writing to Heal course — During this 6-week class, a writing-to-heal instructor will coach participants through a simple progression of writing exercises. Participation requires neither any prior writing experience nor any aspiration to become a writer. In fact, the practices cultivate participants' natural abilities to express the ideas that define who they are and how they experience their lives.
  Weekly sessions build on previous sessions to provide a progression of experiences for participants to develop their natural styles of writing-to-heal. The instructor will guide participants through a variety of modes of writing that enhance health in different ways.

SUMMARY:
The purpose of this study is to determine whether a 6-week writing to heal seminar/workshop/class, Transform Your Life: Write to Heal, raises resilience scores as measured by the Connor-Davidson Resilience Scale for people who have recently experienced an emotional or physical trauma.

Eligible subjects will be adults who self-identify as having had a recent emotional upheaval or physical health challenge. Potential subjects will be recruited through the use of flyers, advertisements, and emails to the Duke Integrative Medicine email list. Subjects will complete pen and paper measures at baseline and immediately post-treatment, including: the Connor-Davidson Resilience Scale, the 10-item Perceived Stress Scale, The 20-item Center for Epidemiological Studies Depression Scale, the 22-item Rumination Response Scale, and a baseline questionnaire.

The investigators aim to target a sample of 30 completers by enrolling 37 participants. The risks of participation in this study are minimal, and include temporary sadness after the initial writing experience.

DETAILED DESCRIPTION:
Background The literature of several health care professions suggests that for many people, writing to heal is beneficial and useful for obtaining and sustaining emotional, physical, and spiritual health. Since the 1980s, a growing body of research shows that the heart rate lowers and people are more equipped to fight off infections when they release their worries in writing. In addition to demonstrating better coping with stressful situations, this research shows that writing can have a positive impact on self-esteem and result in helping people overcome their own obstacles.

Much of the research about writing and healing was pioneered by James Pennebaker, Ph.D., and is now sustained by others who work in the disciplines of writing, psychology, medicine, counseling, nursing, coaching, hospice and education. The biological underpinnings of writing for health are currently found in overlapping scientific areas such as: applied psychoneuorimmunology, psychobiology, applied psychophysiology and recent findings in epigenetics. Research about writing to heal, the kind of writing that is deeply personal and is written for one's own eyes only, demonstrates that such expressive writing:

* Boosts thinking ability
* Increases working memory
* Reduces pain, tension, and fatigue
* Enhances mood and sleep quality
* Positively influences immune system function

Rationale A recent study suggests that writing to heal as part of a larger program may be useful in raising resilience for critical care nurses who have been shown to have lower than average resilience scores on the Connor-Davidson Resilience Scale (2014 Mealer, et.al). In Mealer's multi-modal study, subjects participated in a four hour writing to heal workshop and then wrote according to prescribed prompts once a week for the next twelve weeks. Subjects also participated in Mindfulness-Based Stress Reduction (MBSR) and an exercise program. Post-treatment scores on the CD Resilience Scale were higher for nearly all subjects in this study. However, the potential effect of the writing treatment alone is unclear. Therefore, the aim of this study is to isolate the effect of expressive writing on resilience among those who have experienced an emotional upheaval or a physical health challenge.

Objective: Obtain preliminary data that can be used for grant application addressing the following research question:

Does a 6-week writing to heal workshop, Transform Your Health: Write to Heal, raise resilience, as measured by the Connor-Davidson Resilience Scale for people who have experienced an emotional or physical trauma in the past 12 months?

Design This prospective, observational trial will examine the impact of the 6-week writing course on resilience scores as measured by the Connor-Davidson Resilience Scale (CD-Risc) in a 30-participant pilot trial.

Procedures Potential subjects will be recruited through the use of flyers, advertisements, and via emails to the Duke Integrative Medicine email list.

Potential subjects who call in response to the flyers or who express interest in the study via email will be contacted and screened over the phone by the study coordinator.

Potential subjects will be considered eligible if:

1. They are at least 18 years of age.
2. They self-identify as having had a recent emotional upheaval or physical health challenge (within the past 12 months, but not within the past month).

   a. Potential challenges include, but are not limited to: i. Death of spouse ii. Divorce iii. Marital separation iv. Death of a parent v. Job loss vi. Personal injury or critical illness vii. Death of a close personal friend viii. Retirement ix. Marriage x. Significant change in financial security
3. They are able to read and write in English.
4. They are able to attend 6 weekly sessions of the Transform Your Health: Write to Heal course held at Duke Integrative Medicine.
5. They are able and willing to provide informed consent. The Transform Your Health: Write to Heal course for this study will be devoted entirely to research subjects, and will not be open to the general public.

A group informed consent will be administered by Duke Integrative Medicine staff (either the study coordinator or the principal investigator) during the first session of the course, before any study activities take place. Subjects will do baseline measures (baseline questionnaire, the Connor-Davidson Resilience scale, perceived stress scale, & rumination scale) immediately after the consent.

The expected duration of the subjects' participation is 2 hours each week for 6 weeks, with the first and final classes being slightly longer. The first class in the series will be 2 hours and 30 minutes to allow time for the consent and baseline measures, and the final class will be 2 hours and 30 minutes to allow subjects time to take the post-treatment measures.

In order to have 30 evaluable subjects, using a typical 20% attrition rate for behavioral intervention studies, we plan to consent 37 subjects.

Measures Pen and paper measures will be collected at baseline and immediately post-treatment.

Primary outcome:

1. Connor-Davidson Resilience Scale (CD-RISC): This 25-item scale addresses resilience, and has been studied in a variety of populations. Resilience is considered as the capacity to overcome adversity.

Secondary measures:

1. Baseline questionnaire: This self-report questionnaire will gather basic sociodemographic information (i.e., gender, age, ethnicity, race, marital status, living situation, education). This questionnaire will be given at baseline only.
2. 10-item Perceived Stress Scale (PSS-10): The PSS a well-known 10-item questionnaire used to evaluate responders' perceptions about their level of stress and their ability to cope with stress over the last month. Results from this questionnaire have demonstrated acceptable levels of validity and reliability. This inventory asks participants to respond using a 10-point Likert-type scale when endorsing the degree to which each item best reflects their thoughts and feelings within the past month (Cohen, Kamarck, & Mermelstein, 1983).
3. 20-item Center for Epidemiological Studies Depression Scale (CES-D): The CES-D is one of the most common screening tests that measures depressive feelings and behaviors within the past week. Almost 85% of those found to have depression after an in-depth structured interview with a psychiatrist will have a high score on the CES-D. However, about 20% of those who score high on the CES-D will have rapid resolution of their symptoms and not meet full criteria for major or clinical depression (Radloff, 1977).
4. 22-item Rumination Response Scale (RRS): The RRS is questionnaire used to examine response styles for depression (Nolen-Hoeksema, 2003).

Compensation Subjects will receive the 6-week Transform Your Health: Write to Heal class at no cost. There is no monetary compensation for this study.

Curriculum During this 6-week class, an experienced writing-to-heal instructor will coach participants through a simple progression of writing exercises. Participation requires neither any prior writing experience nor any aspiration to become a writer. In fact, the practices cultivate participants' natural abilities to express the ideas that define who they are and how they experience their lives.

Weekly sessions build on previous sessions to provide a progression of experiences for participants to develop their natural styles of writing-to-heal. The instructor will guide participants through a variety of modes of writing that enhance health in different ways, including:

i. Expressive Writing: moving beyond what you thought you could not get over. ii. Transactional Writing: communicating your desires with compassion, empathy, forgiveness and gratitude.

iii. Poetic Writing: expressing your "rites of passage" with metaphor, story, poetry and creative nonfiction.

iv. Affirmative Writing: discovering your gifts and describing your best possible life by writing it forward.

v. Legacy Writing: sharing your values and the life lessons you have learned for those you love.

Data Analysis & Statistical Considerations Given that the objective is to obtain pilot data for a future grant, we will target a sample of 30 completers by enrolling 37 participants. Relying on the tenets of the Central Limit Theorem and how scores on CD-RISC have behaved in other trials, we expect to have a fairly normal distribution of scores at both time points that will allow a simple dependent-measures t-test to estimate any change from pre to post intervention.

Discomforts and Risks The risks of participation in this study are minimal. Participants may experience a range of emotions, including sadness after the initial expressive writing experience. This is a common occurrence in this course and sadness is usually brief before negative mood lifts.

Potential Benefits Some participants who have taken the course have reported physical and emotional benefits, including a more balanced mood, increased ability to sleep, lower blood pressure, fewer symptoms of depression (Pennebaker & Evans, 2014; Stockdale, 2011).

Confidentiality Every effort will be made to keep participants' information confidential. Subject study records will be assigned a unique code number, and the key to this code will be kept in a password-protected computer file in the principal investigator's or study coordinator's office until the completion of the study. All consent forms and questionnaire information will be stored separately in a locked file drawer in the study coordinator's office. All data considered sensitive electronic information will be stored on a DHTS network drive.

Additionally, participants' personal writing is not required to be shared and responses to the writing remain anonymous.

ELIGIBILITY:
Inclusion Criteria:

1. They are at least 18 years of age.
2. They self-identify as having had a recent emotional upheaval or physical health challenge (within the past 12 months, but not within the past month).

   a. Potential challenges include, but are not limited to: i. Death of spouse ii. Divorce iii. Marital separation iv. Death of a parent v. Job loss vi. Personal injury or critical illness vii. Death of a close personal friend viii. Retirement ix. Marriage x. Significant change in financial security
3. They are able to read and write in English.
4. They are able to attend 6 weekly sessions of the Transform Your Health: Write to Heal course held at Duke Integrative Medicine.
5. They are able and willing to provide informed consent.

Exclusion Criteria:

1. They are NOT at least 18 years of age.
2. They do NOT self-identify as having had a recent emotional upheaval or physical health challenge (within the past 12 months, but not within the past month).
3. They are NOT able to read and write in English.
4. They are NOT able to attend 6 weekly sessions of the Transform Your Health: Write to Heal course held at Duke Integrative Medicine.
5. They are NOT able and willing to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Connor-Davidson Resilience Scale (CD-RISC) | 6 weeks

SECONDARY OUTCOMES:
10-Item Perceived Stress Scale (PSS-10) | 6 weeks
20-item Center for Epidemiological Studies Depression Scale (CES-D) | 6 weeks
22-item Rumination Response Scale (RRS) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adam Perlman, MD, Principal Investigator — Duke University
Locations (1):
- Duke Integrative Medicine, Durham, North Carolina, United States